CLINICAL TRIAL: NCT02866435
Title: Identifying the Brain Substrates of Hypoglycemia Unawareness in Type 1 Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1608M92941
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Hypoglycemia
Keywords: MRI
MeSH Terms: conditions — Hypoglycemia | interventions — Insulin; Insulin, Regular, Human; Glucose; potassium phosphate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Euglycemia pre-conditioning (Experimental): Participants will undergo two euglycemia (normal blood sugar) clamps (8-10 am and 1-3 pm) on day 1, where the target glucose during the clamp will be 95 mg/dl. For each clamp, participants will be given intravenous insulin for two hours and blood glucose will be maintained at target by the infusion of 20% dextrose, the rate of which will be adjusted based on measured blood glucose values collected every 5 minutes. Potassium phosphate will also be infused during each clamp. On next day (day 2), participants will undergo MRI session during experimental hypoglycemia, i.e., while their blood sugar is clamped from normal value to low value.
  Interventions: Drug: Insulin; Drug: Glucose; Drug: Potassium phosphate
- Hypoglycemia pre-conditioning (Experimental): Participants will undergo two hypoglycemia (low blood sugar) clamps (8-10 am and 1-3 pm) on day 1, where target glucose during the clamp will be 50 mg/dl. For each clamp, participants will be given intravenous insulin for two hours and blood glucose will be maintained at target by the infusion of 20% dextrose, the rate of which will be adjusted based on measured blood glucose values collected every 5 minutes. Potassium phosphate will also be infused during each clamp. On next day (day 2), participants will undergo MRI session during experimental hypoglycemia, i.e., while their blood sugar is clamped from normal value to low value.
  Interventions: Drug: Insulin; Drug: Glucose; Drug: Potassium phosphate

INTERVENTIONS:
Drug: Insulin — In each clamp, a small intravenous catheter is placed in participant's arm for infusion of insulin together with potassium phosphate and glucose. Insulin is a hormone that body makes naturally and it causes blood sugar to decrease. Insulin (and glucose) will be infused in calculated doses to maintain blood sugar level in the target range of 95 mg/dl or 50 mg/dl depending on the clamp.
  Other Names: Humulin
Drug: Glucose — Glucose is administered together with insulin and potassium phosphate during each clamp via the intravenous catheter. Glucose is a sugar and it is used to carefully regulate blood sugar level.
  Other Names: Dextrose
Drug: Potassium phosphate — Potassium phosphate is administered together with glucose and insulin during each clamp via the intravenous catheter. Potassium is a salt-like substance that is present in the blood.
  Other Names: K Phos

SUMMARY:
The purpose of this study is to investigate how the brain responds to low blood glucose in non-diabetic individuals. The ultimate goal is to understand the brain substrates of hypoglycemia unawareness, a condition that can occur in patients with type1 diabetes undergoing insulin treatment.In the present study, the investigators focus on differences between two groups of non-diabetic subjects: one group who experienced two episodes of hypoglycemia the day prior to the study (and supposedly developed some level of unawareness to hypoglycemia), and one group who did not. In this study, a 3 tesla MRI scanner is used to acquire brain images. The imaging system is identical to the ones used in hospitals.

DETAILED DESCRIPTION:
Hypoglycemia, also called low blood glucose or low blood sugar, occurs when blood glucose drops below normal levels. When blood glucose starts to drop, the body reacts to this drop, trying to restore the blood glucose level. Symptoms of hypoglycemia are usually easily recognized. Hypoglycemia can be treated quickly and easily by eating or drinking a small amount of glucose-rich food. However some people with long history of diabetes can have an impaired response to hypoglycemia and therefore don't recognize the symptoms of hypoglycemia, condition called hypoglycemia unawareness. If not treated hypoglycemia can get worse and cause confusion, clumsiness, fainting etc. Currently, it is not fully understood which brain areas are involved in sensing the drop of glucose levels. Absence of such knowledge is a critical barrier to the design and monitoring of effective intervention strategies to avoid and/or reverse hypoglycemia unawareness. The purpose of this study is to investigate how the brain responds to low blood glucose in non-diabetic individuals. Specific focus is given to differences between two groups of non-diabetic subjects: one group who experienced two episodes of hypoglycemia the day prior to the study (and therefore supposedly developed some level of unawareness to hypoglycemia), and one group who did not.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included in the study, if they

* are non-diabetic
* are evaluated as not contraindicated (based on exclusion criteria)
* are age (within 5 years), gender, and body mass index (within 4 kg/m2) matched to patients with type 1 diabetes who have participated to a similar study which involved only the second part (day 2) of the current protocol.

Exclusion Criteria:

Participants will be excluded from the study, if they

* have any type of bio-implant activated by mechanical, electronic, or magnetic means (e.g. cochlear implants, pacemakers, neurostimulators, bio stimulators, electronic infusion pumps)
* have any type of ferromagnetic bio-implant that could potentially be displaced or damaged, such as aneurysm clips, metallic skull plates, etc
* have any retained metal in their body, either from a medical procedure or an injury
* have history of stroke, seizures, neurosurgical procedures, or arrhythmias
* are pregnant
* are currently using medication that can alter glucose metabolism or brain perfusion
* weight more than 300lbs (limit for MRI scanner)
* have concomitant medical problems that may prevent them from successfully completing the protocol
* lack capacity to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline (i.e., normal glucose levels) functional connectivity, measured as a dimensionless correlation coefficient of MRI signals among brain areas, at hypoglycemia | Baseline and immediately as hypoglycemia starts
  Functional connectivity will be measured with MRI at 3 Tesla
Change from baseline (i.e., normal glucose levels) cerebral blood flow, measured in ml/min/100g, at hypoglycemia | Baseline and immediately as hypoglycemia starts
  Cerebral blood flow will be measured with MRI at 3 Tesla

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Mangia, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mangia S, Tesfaye N, De Martino F, Kumar AF, Kollasch P, Moheet AA, Eberly LE, Seaquist ER. Hypoglycemia-induced increases in thalamic cerebral blood flow are blunted in subjects with type 1 diabetes and hypoglycemia unawareness. J Cereb Blood Flow Metab. 2012 Nov;32(11):2084-90. doi: 10.1038/jcbfm.2012.117. Epub 2012 Aug 15. PMID 22892724
- [Background] Bolo NR, Musen G, Simonson DC, Nickerson LD, Flores VL, Siracusa T, Hager B, Lyoo IK, Renshaw PF, Jacobson AM. Functional Connectivity of Insula, Basal Ganglia, and Prefrontal Executive Control Networks during Hypoglycemia in Type 1 Diabetes. J Neurosci. 2015 Aug 5;35(31):11012-23. doi: 10.1523/JNEUROSCI.0319-15.2015. PMID 26245963
- [Background] Wiegers EC, Becker KM, Rooijackers HM, von Samson-Himmelstjerna FC, Tack CJ, Heerschap A, de Galan BE, van der Graaf M. Cerebral blood flow response to hypoglycemia is altered in patients with type 1 diabetes and impaired awareness of hypoglycemia. J Cereb Blood Flow Metab. 2017 Jun;37(6):1994-2001. doi: 10.1177/0271678X16658914. Epub 2016 Jan 1. PMID 27389175
- [Background] Rooijackers HM, Wiegers EC, Tack CJ, van der Graaf M, de Galan BE. Brain glucose metabolism during hypoglycemia in type 1 diabetes: insights from functional and metabolic neuroimaging studies. Cell Mol Life Sci. 2016 Feb;73(4):705-22. doi: 10.1007/s00018-015-2079-8. Epub 2015 Oct 31. PMID 26521082
- See also: Description Profile of Principal Investigator — http://www.cmrr.umn.edu/facultystaff/mangia/